CLINICAL TRIAL: NCT06708845
Title: A Phase I Multicohort Trial of Zamtocabtagene Autoleucel (Zamto-Cel) in Subjects with Severe Refractory Autoimmune Diseases
Brief Title: US Zamto-cel Autoimmune Diseases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M-2024-423
Record Dates: First submitted 2024-11-26; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Lupus Nephritis; Systemic Lupus Erythematosus; Systemic Sclerosis (SSc); Diffuse Cutaneous Systemic Sclerosis
Keywords: Chimeric antigen receptor; CAR T; Zamtocabtagene autoleucel; Autoimmune Disease; Immune System Diseases; SLE-Non renal; SLE-LN; SSc; dcSSc; Lupus
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Scleroderma, Diffuse; Autoimmune Diseases; Immune System Diseases | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Level 1 (Experimental)
  Interventions: Biological: zamtocabtagene autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Dose Level 2 (Experimental)
  Interventions: Biological: zamtocabtagene autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: zamtocabtagene autoleucel — chimeric antigen receptor T-cell (CAR-T) therapy
Drug: Cyclophosphamide — Lymphodepleting chemotherapy
Drug: Fludarabine — Lymphodepleting chemotherapy

SUMMARY:
AID is a phase I multi-cohort study to assess the safety and tolerability of zamtocabtagene autoleucel (zamto-cel) in patients with refractory autoimmune diseases (SLE-Non renal, SLE-LN, SSc/dcSSc) after receiving standard therapy.

DETAILED DESCRIPTION:
This is a Phase 1, multicohort, dose-finding study evaluating autologous T cells engineered to target dual CD19 and CD20 antigens in subjects with refractory autoimmune diseases following standard therapy. The investigational product, Zamto-cel, is a chimeric antigen receptor T-cell (CAR-T) therapy genetically engineered to enable subjects' T cells to express CARs on their surfaces.

Eligible subjects will undergo leukapheresis for the collection of cells required for manufacturing. Prior to infusion of the fresh CAR-T product, subjects will receive a lymphodepleting regimen consisting of cyclophosphamide and fludarabine. The CAR-T cell infusion will be administered intravenously at a dose of 2.5 x 10^6 or 1.0 x 10^6 CAR+ cells/kg body weight, based on the dose level assigned to the cohort.

The study will initially enroll 3 subjects per cohort in a staggered manner to evaluate safety. Upon confirmation of safety, the study will proceed to cohort-specific recommended Phase 2 dose (RP2D) and dose expansion phases. Subjects will be monitored for up to 1 year to assess safety, preliminary efficacy, and health-related quality of life (HRQoL). Additional long-term follow-up will be conducted under a separate long-term follow-up protocol.

ELIGIBILITY:
General Key Inclusion/Exclusion Criteria Across All Cohorts

Inclusion Criteria:

•Confirmed diagnosis of autoimmune disease (SLE-Non-renal, SLE-LN, SSc/ dcSSc)

Exclusion Criteria:

* Prior gene therapy treatment
* Active malignancy within past 5 years
* Significant active fungal or bacterial infection
* History or presence of CNS lupus or other CNS disease
* eGFR < 45 mL/min/1.73 m^2
* Total bilirubin outside the normal range (unless congenital hyperbilirubinemia such as Gilbert syndrome has been confirmed).

Systemic Lupus Erythematosus-Non-renal Key Inclusion/Exclusion Criteria

Inclusion Criteria:

* Positive for at least 1 of the following autoantibodies at Screening: anti- double stranded DNA or anti-Smith
* Systemic Lupus Erythematosus Disease Activity Index-2000 score ≥ 8 AND at least 1 British Isles Lupus Assessment Group (BILAG)-2004 Class A (severe manifestation) organ scores
* Inadequate response to glucocorticoids and to at least 2 of the following treatments, used for at least 3 months each: cyclophosphamide, mycophenolic acid or its derivatives, belimumab, azathioprine, anifrolumab, methotrexate, rituximab, or obinutuzumab

Exclusion Criteria:

* Subjects with neuropsychiatric SLE.
* Drug-induced SLE.

Systemic Lupus Erythematosus - Lupus Nephritis Key Inclusion/Exclusion Criteria

Inclusion Criteria:

* Positive for at least 1 of the following autoantibodies at Screening: anti- double stranded DNA or anti-Smith
* Confirmed LN diagnosis by kidney biopsy during screening or within the previous 6 months, with severe active phase of the disease.
* Progressing despite maintenance on maximally tolerated doses of renin- angiotensin system (RAS) blocking agents, unless allergic to or intolerant of ACE inhibitors and ARBs
* Inadequate response to glucocorticoids and hydroxychloroquine and at least 1 of the following treatments, used for at least 3 months each: cyclophosphamide, mycophenolic acid derivatives, belimumab, azathioprine, methotrexate, rituximab, obinutuzumab, calcineurin inhibitor (cyclosporin, tacrolimus or voclosporin)

Exclusion Criteria:

•Evidence of Rapidly progressive glomerulonephritis (defined as a doubling of serum creatinine within 3 months prior to enrollment) or as determined by the study investigator.

Systemic Sclerosis/Diffuse Cutaneous Systemic Sclerosis Cohort Key Inclusion/ Exclusion Criteria

Inclusion Criteria:

* Active disease defined as:
* Modified Rodnan skin score (mRSS) ≥ 16 units, in the prior 6 months, with 1 or more of the following:

  * Increase in mRSS by ≥ 3 units or 10%
  * Involvement of 1 new body area with increase in mRSS by ≥ 2 units
  * Involvement of 2 new body areas with increase by ≥ 1 mRSS unit OR
* Progressive interstitial lung disease (ILD) defined as:

  - Worsening of respiratory symptoms and an increased extent of fibrosis evaluated by high-resolution computed tomography
* Lack of response to standard therapy (e.g., failure of ≥ 2 immunosuppressive therapies)

Exclusion Criteria:

* "Active" gastric antral vascular ectasia, as evidenced by bleeding (ie, on esophagogastroduodenoscopy) in the past 6 months or as per Investigator's assessment.
* History of SSc renal crisis within 1 year prior to Screening; presence of kidney impairment due to conditions other than SSc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events (AEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) | From enrollment through study completion 12 months post zamto-cel infusion
The proportion of subjects with dose-limiting toxicities (DLTs) up to Day 28 and determination of recommended Phase 2 dose (RP2D) | From enrollment through Day 28 post zamto-cel infusion

SECONDARY OUTCOMES:
The incidence and severity of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) | From enrollment through study completion 12 months post zamto-cel infusion
Clinical response at Week 4, 12, 24, and 52 evaluated by defined disease-specific activity measures in SLE-Non renal, SLE-LN, and SSc/dcSSc | From enrollment through study completion 12 months post zamto-cel infusion
The duration of remission or low disease activity status in respective diseases under the study | From enrollment through study completion 12 months post zamto-cel infusion
Persistence, maximal drug concentration (Cmax), time to reach Cmax, area under the concentration curve, and phenotype of zamto-cel | From enrollment through study completion 12 months post zamto-cel infusion

CONTACTS AND LOCATIONS:
Overall Officials: Esther Eromosele, MD, Study Director — Miltenyi Biomedicine

IPD SHARING:
Plan to Share IPD: No